CLINICAL TRIAL: NCT00224991
Title: Effect of Training in Prevention of Falls, Compliance to Treatment and Quality of Life: A Randomized, Prospective Investigation.
Brief Title: Osteoporosis School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: ON-06-001-AJ
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Osteoporosis
Keywords: osteoporosis; fall frequency; medical treatment; compliance; quality of life; systematic education
MeSH Terms: conditions — Osteoporosis; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Intensive systematic information (osteoporosis school)

SUMMARY:
The purpose of this study is to investigate the efficacy of systematic education (osteoporosis school) on fall frequency, compliance and quality of life of a group of patients more than fifty years of age.

Hypothetically, systematic information can increase compliance to the medical treatment, decrease the frequency of falls and increase the quality of life.

DETAILED DESCRIPTION:
In most randomized trials compliance to medical treatment in osteoporosis is very high, but compliance tends to be considerably inferior in routine treatment compared to scientific trials. This fact is caused by a narrow selection of motivated patients in the randomized trials. Perhaps, the information given to the patients in scientific trials is more thorough than information given in a routine setting.

There are no trials available that document that compliance to medical treatment of patients with osteoporosis can be increased by intensive systematic information.

Change of lifestyle is an important part in the treatment of these patients. The patients are encouraged to eat more healthy food combined with an intake of calcium and vitamins, reduction of alcohol and tobacco consumption if needed and prevention of fall incidence through changes in the house.

The quality of life is often reduced, partly due to chronic pain, altered social status, physical handicap and partly due to the heavy knowledge of having a chronic decease.

Adaption to the last-mentioned factors can possibly lead to a considerably better quality of life in spite of the unchanged physical handicap.

Randomized trials on efficacy of systematic patient education has in general been positive in other contexts. Young patients with diabetes offered coping skills training have therefore a better metabolic control and quality of life.

No similar randomized trials are available on the efficacy of a systematic education program in osteoporosis.

ELIGIBILITY:
Inclusion criteria:

* fracture caused by osteoporosis
* fifty years or more of age
* informed consent

Exclusion criteria:

- Physically or mental state that does not participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 1999-06; Study Completion 2005-06

PRIMARY OUTCOMES:
Fall frequency

SECONDARY OUTCOMES:
Compliance
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Annette Jaquet, Principal Investigator — Northern Orthopaedic Division
Locations (1):
- Northern Orthopaedic Division, Klinik Hjoerring, Hjørring, Northern Jutland, Denmark